CLINICAL TRIAL: NCT02136732
Title: Chronic Care Management Model Translation to Multimorbid Aging Adults at FQHCs
Brief Title: Chronic Care Management for Adults at FQHCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington State University (Other)
Collaborators: Community Health Association of Spokane (Unknown); Aging and Long Term Care of Eastern Washington (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01AG042467-01A1 (NIH)
Record Dates: First submitted 2013-11-07; First posted 2014-05-13 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Any Condition in N73.0 Specified as Chronic
Keywords: chronic conditions; multimorbid
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active self-management intervention (Experimental): Participants will receive home visits and phone calls from a registered nurse and social worker. The registered nurse and social worker will provide participants one on one coaching, education, support and referrals to community resources to help them manage their chronic conditions.
  Interventions: Other: Active self-management intervention
- Attention control phone calls (Active Comparator): Participants will receive an initial visit and then a phone call every other month from a social services aide who can provide information about community resources that might be helpful.
  Interventions: Other: Attention control phone calls

INTERVENTIONS:
Other: Active self-management intervention — Participants will set health goals at baseline. They will then receive, at minimum, a visit or a phone call to assess how progress and coaching toward meeting goals on a monthly basis from a nurse and/or social worker. The frequency and exact activities associated with the intervention are dependent on each participant's unique health goals.
  Arms: Active self-management intervention
Other: Attention control phone calls — Participants will be called by a social service aide at 2, 4, 6, 8, 10, and 12 months.
  Arms: Attention control phone calls

SUMMARY:
With a growing aging population, the number of persons with chronic conditions continues to escalate and challenges related to chronic care quality, effectiveness and cost remain unresolved.Federally Qualified Health Centers (FQHC) have experienced increasing numbers of patient visits for chronic conditions, and FQHC patients are more likely to have serious chronic conditions when compared to patients being cared for by non-FQHC providers.

The Chronic Care Intervention (CCI) combines home visiting with health activation coaching and has resulted in improved health status and reduced expenditures (Preliminary Studies). Implementing the CCI for aging adults with multimorbidity (2 or more chronic conditions) and high baseline acute care utilization, allows us to test and expand the efficacy, external validity and cost effectiveness of the proposed intervention model. The investigators seek to improve patients' and FQHCs' abilities to effectively manage chronic conditions and reduce acute care use. This contribution is significant because it potentially extends our knowledge about effective community partnerships and best practices that can enhance the effectiveness of health homes in providing patient-centered team-based care for patients with multimorbidity and high baseline health care utilization.

DETAILED DESCRIPTION:
With a growing aging population, the number of persons with chronic conditions continues to escalate and challenges related to chronic care quality, effectiveness and cost remain unresolved. Federally Qualified Health Centers (FQHC) have experienced increasing numbers of patient visits for chronic conditions, and FQHC patients are more likely to have serious chronic conditions when compared to patients being cared for by non-FQHC providers. Effectively managing multiple chronic conditions is particularly challenging for both patients and health professionals, and costs of care rise as the number of co-morbid conditions increases. FQHCs primarily serve patients with public insurance or those who are uninsured. Consequently, simultaneously controlling costs and improving chronic care is a critical issue for the FQHC system. Two approaches that have been used to improve health status and reduce health care utilization are preventive home visiting and patient activation counseling. Preventive home visiting allows for multidimensional assessment and individualized, patient-centered care, and there is wide agreement that engaging patients to be an active part of the care process is an essential element of the quality of care. This concept is known as "health activation".

The Chronic Care Intervention (CCI) combines home visiting with health activation coaching and has resulted in improved health status and reduced expenditures (Preliminary Studies). Implementing the CCI for aging adults with multimorbidity (2 or more chronic conditions) and high baseline acute care utilization, allows us to test and expand the efficacy, external validity and cost effectiveness of the proposed intervention model. The investigators seek to improve patients' and FQHCs' abilities to effectively manage chronic conditions and reduce acute care use. This contribution is significant because it potentially extends our knowledge about effective community partnerships and best practices that can enhance the effectiveness of health homes in providing patient-centered team-based care for patients with multimorbidity and high baseline health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older, 2 or more chronic conditions, 2 or more emergency department visits or hospital admissions in previous 12 months.

Exclusion Criteria:

* terminal illness, dementia, case management elsewhere, resident of adult family home, boarding home or skilled nursing facility, homeless.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
patient activation | change from baseline to 3, 6, and 12 months
  Patient activation will be measured using the Patient Activation Measure. Higher scores on this tool indicate that the patient is more involved in self-managing care and partnering with health care professionals to achieve better health outcomes.

SECONDARY OUTCOMES:
acute care utilization | change in acute care utilization from baseline year to intervention year
  Acute care utilization is defined as visits to the emergency department and admissions to the hospital

OTHER OUTCOMES:
Participant's Health-Related Quality of Life. | change in quality of life from baseline to 3 months, 6 months, 9 months, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Corbett, Ph.D., Principal Investigator — Washington State University College of Nursing
Locations (1):
- Community Health Association of Spokane, Spokane, Washington, United States